CLINICAL TRIAL: NCT04875260
Title: Taiwan Center of Outcome and Resource Evaluation Adult Intensive Care Units Database
Brief Title: Taiwan Center of Outcome and Resource Evaluation
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006006RINA
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Patients received critical care in the intensive care units
  Interventions: Other: Critical Care

INTERVENTIONS:
Other: Critical Care — Critical care in the intensive care units

SUMMARY:
The main purpose of this proposal is to build a multicenter de-identification adult intensive care units database in Taiwan. In future, the Joint Data Management Committee and investigators can use the data for evaluation of outcome of critical care, evaluation of medical resource, quality improvement, annual report, education and training, and critical care research.

Center of Outcome and Resource Evaluation (CORE) Adult Patient Database of Australian and New Zealand Intensive Care Society (ANZICS) was founded in 1992. More than 160 intensive care units in Australia and New Zealand contribute the data into this database. This database provides medical information to Australia and New Zealand government for critical care policy making and quality improvement. The primary aim of this proposal is to build a multicenter de-identification adult intensive care units database by mutual collaboration of multiple hospitals in Taiwan. This database will include the de-identification data accruing to the regulation of Health Insurance Portability and Accountability Act (HIPAA) of United States of America from each hospital. The data can be used to help the government and critical care societies evaluate the clinical outcomes of critical care. Furthermore, this data can help to effectively allocate the medical resource, improve quality, conduct multicenter registry-based clinical research, and publish high quality research. Hope to assist Taiwan and the world to improve critical care quality.

DETAILED DESCRIPTION:
The main purpose of this proposal is to build a multicenter de-identification adult intensive care units database in Taiwan. In future, the Joint Data Management Committee and investigators can use the data for evaluation of outcome of critical care, evaluation of medical resource, quality improvement, annual report, education and training, and critical care research.

Center of Outcome and Resource Evaluation (CORE) Adult Patient Database of Australian and New Zealand Intensive Care Society (ANZICS) was founded in 1992. More than 160 intensive care units in Australia and New Zealand contribute the data into this database. This database provides medical information to Australia and New Zealand government for critical care policy making and quality improvement. The primary aim of this proposal is to build a multicenter de-identification adult intensive care units database by mutual collaboration of multiple hospitals in Taiwan. This database will include the de-identification data accruing to the regulation of Health Insurance Portability and Accountability Act (HIPAA) of United States of America from each hospital. The data can be used to help the government and critical care societies evaluate the clinical outcomes of critical care. Furthermore, this data can help to effectively allocate the medical resource, improve quality, conduct multicenter registry-based clinical research, and publish high quality research. Hope to assist Taiwan and the world to improve critical care quality.

The Taiwan Society of Critical Care Medicine, Taiwan Society of Emergency and Critical Care Medicine, and National Taiwan University Hospital invite multiple hospitals to build the multicenter de-identification adult intensive care units database. This database includes only de-identification data. A Joint Data Management Committee will be organized and be in charge of data management. The data will be used for evaluation of outcome of critical care, evaluation of medical resource, quality improvement, and publication of mutual collaboration of critical care research in research ethic committee approved research filed.

ELIGIBILITY:
Inclusion Criteria:

* •Critically ill patients admitted to intensive care units

Exclusion Criteria:

* •Critically ill patients admitted to intensive care units

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 600000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2040-07 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  mortality status at 30 days after admission to intensive care unit

SECONDARY OUTCOMES:
Length of stay in intensive care units | a median 2 to 7 days
  Number of days in intensive care unite

CONTACTS AND LOCATIONS:
Locations (10):
- Taiwan (10):
  - National Taiwan University Hospital Yun-Lin Branch, Douliu
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veteran General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Medical Foundation, Taoyuan District